CLINICAL TRIAL: NCT01612065
Title: The Optimum Dose of Vaginal Misoprostol Prior to Office Hysteroscopy: Double Blind Randomized Controlled Trial
Brief Title: Optimum Misoprostol Dose Prior to Office Hysteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assistant professor of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2752012
Record Dates: First submitted 2012-05-28; First posted 2012-06-05 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Infertility; Abnormal Uterine and Vaginal Bleeding, Unspecified; Recurrent Abortion
Keywords: Office hysteroscopy; Cervical priming; Misoprostol
MeSH Terms: conditions — Infertility; Uterine Hemorrhage; Abortion, Habitual | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Misoprostol vaginally, 200 ug (Active Comparator): 200 ug misoprostol in the posterior vaginal fornix
  Interventions: Drug: Misoprostol
- Misoprostol vaginally, 400ug (Active Comparator): Misoprostol in the posterior vaginal fornix
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 200 ug
  Arms: Misoprostol vaginally, 200 ug
Drug: Misoprostol — Misoprostol vaginally, 400 ug
  Arms: Misoprostol vaginally, 400ug

SUMMARY:
Misoprostol is an effective agent for cervical priming before office hysteroscopy, vaginal route is the best, optimum dose not yet known.

DETAILED DESCRIPTION:
The investigators will compare between 2 different doses of vaginal misoprostol, group (1) 200 ug, group (2) 400 ug, 3hours prior to office hysteroscopy , Infertile patient, patients with abnormal bleeding and patient with recurrent abortion Outcome measure: pain score, easiness of the procedure, procedure time, complications

ELIGIBILITY:
Inclusion Criteria:

* Female patient pre- or postmenopausal undergo office hysteroscopy.
* Age: from 20 to 60.
* BMI between 18 and 30.

Exclusion Criteria:

* PID or
* Heavy uterine bleeding
* Cervical malignancy.
* Symptoms suggestive of endometriosis .
* Any cervical abnormality such as pinhole cervix that would obviate passage of a catheter through the cervix.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain score | 1year
  Pain score by VAS

SECONDARY OUTCOMES:
Easiness | 1year
  ease of entry of the office hysteroscopy into the cervix recorded on a 5-point Likert scale: very difficult= 1, difficult = 2, fair = 3, easy = 4, and very easy = 5;
Duration of the procedure | 1year
  Duration of hysteroscopy in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khayat, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr alainy hospital, faculty of medicine , Cairo university, Cairo, Egypt